CLINICAL TRIAL: NCT05512832
Title: Construction and Evaluation of Clinical Prediction Model of In-stent Restenosis After Percutaneous Coronary Intervention by Pericoronary Fat Attenuation Index and Radiomics Characteristics
Brief Title: In-stent Restenosis and Pericoronary Fat Attenuation Index
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: EARLY-ISR FAI
Record Dates: First submitted 2022-08-17; First posted 2022-08-23 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: In-stent Restenosis
Keywords: pericoronary fat attenuation index

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ISR: Patient developed in-stent restenosis 9-24 months after stenting
- no ISR: Patients were free of in-stent restenosis 9-24 months after stenting

SUMMARY:
This study aims to investigate the predictive value of fat attenuation index (FAI) and related radiomics characteristics of pericoronary fat in patients after percutaneous coronary intervention (PCI) for the occurrence of in-stent restenosis (ISR) during the follow-up period (9 to 24 months). The results of this study are expected to provide an early assessment of the inflammation around the coronary lesion segment in patients after PCI, and provide a basis for early targeted intensive drug therapy in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with coronary heart disease who have undergone PCI;
* Patients followed up coronary angiography 9 to 24 months after PCI;
* Patients received chest CT examination during inpatient/outpatient follow-up;

Exclusion Criteria:

* Patients with diseases of the immune system;
* Patients with history of tumor diseases;
* Patients with chronic/acute infectious diseases;
* Image quality is not sufficient for analysis;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with coronary heart disease who have undergone PCI and followed up angiography 9 to 24 months after PCI
Sampling Method: Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Fat attenuation index (FAI) | 2022.8.15-2023.8.14
  The pericoronary FAI was defined as the mean CT attenuation of the pericoronary adipose tissue (-190 to -30 HU). Peri-stent FAI was measured around the stent segment of all 3 major epicardial coronary vessels.

CONTACTS AND LOCATIONS:
Overall Officials: Song Ding, Principal Investigator — RenJi Hospital
Locations (1):
- Cardiology, Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No